CLINICAL TRIAL: NCT04741022
Title: The Prevalence and Influence of Obstructive Sleep Apnea in Coronary Artery Disease in Modern Age: Findings in A Large Cohort Study
Brief Title: Influence of Obstructive Sleep Apnea on the Severity of Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Chinese Pulmonary Vascular Disease Research Group (Other)
Responsible Party: Sponsor
Other Study IDs: IOSAC
Record Dates: First submitted 2021-02-03; First posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2019-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CAD with OSA: coronary artery disease with Obstructive sleep apnea
- CAD without OSA: coronary artery disease without Obstructive sleep apnea

SUMMARY:
It is widely accepted that coronary artery disease (CAD) is related to a high mortality. It is predicted that an increase of approximately 21.3 million cardiovascular events and 7.7 million cardiovascular deaths over 2010 to 2030 in China.1 Male sex, diabetes mellitus, hypertension, hypercholesterolemia, obesity and smoking are all traditionally considered as risk factors for CAD. In recent decades, tremendous progress toward the prevention and treatment of traditional cardiovascular risk factors have helped decrease the morbidity and mortality from CAD, but the condition remains a major public health challenge worldwide. Looking into the other potential risk factors (OSA) for CAD, it may help to develop additional preventative strategies and further reduce the incidence and mortality of CAD.

DETAILED DESCRIPTION:
Before initiating the study, all potential subjects were invited to attend an educational program that explained the purpose and methodology of this study. After getting informed consent from patients, demographic data including age, sex, medical history (including comorbidities and risk factors), current medicine, lifestyle habits, height (cm), and weight (kg) were recorded, and body mass index (BMI) was calculated as weight divided by height squared (kilograms per square meter, kg/m2). The included subjects need to perform transthoracic echocardiography or provide an echocardiographic examination within one month. CAD diagnosis was determined based on the results of the coronary angiography, using stenosis 50% cutoffs considered have coronary diseases or not.

Consecutive patients of both sexes with coronary angiography from outpatient or inpatient departments of Fuwai Hospital were recruited into the study. The inclusion criteria were Chinese, aged 35 to 75 years with CAD verified by coronary angiography, and able to give informed written consent. The subjects were excluded if they had New York Heart Association Class III-IV degree with ejection fraction < 45%, severe pulmonary disease, significant psychiatric disease, or history of pharyngeal surgery for OSA or current use of CPAP treatment for OSA. They were also excluded if they declined to participate or were unable to provide informed consent.

ELIGIBILITY:
Inclusion Criteria:

* aged 35 to 75 years with CAD
* CAD was verified by coronary angiography

Exclusion Criteria:

* Patients had New York Heart Association Class III-IV degree with ejection fraction < 45%
* Severe pulmonary disease
* Significant psychiatric disease
* History of pharyngeal surgery for OSA or current use of CPAP treatment for OSA
* Subjects declined to participate or were unable to provide informed consent.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients of both sexes with coronary angiography from outpatient or inpatient departments of Fuwai Hospital were recruited into the study. The inclusion criteria were Chinese, aged 35 to 75 years with CAD verified by coronary angiography, and able to give informed written consent. The subjects were excluded if they had New York Heart Association Class III-IV degree with ejection fraction < 45%, severe pulmonary disease, significant psychiatric disease, or history of pharyngeal surgery for OSA or current use of CPAP treatment for OSA. They were also excluded if they declined to participate or were unable to provide informed consent.
Sampling Method: Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

PRIMARY OUTCOMES:
Association of apnea-hypopnea index (AHI) between obstructive sleep apnea and severity of coronary artery disease | 12 months
  The apnea-hypopnea index (AHI) was calculated as the total number of apneas and hypopneas occurring per hour of sleep. And the severity of coronary artery disease was determined by Coronary angiography.

SECONDARY OUTCOMES:
The Prevalence of Obstructive Sleep Apnea in Coronary Artery Disease in China | 12 months
  The number of patients with Obstructive Sleep Apnea in Coronary Artery Disease in China

CONTACTS AND LOCATIONS:
Overall Officials: Zhihong Liu, M.D, Study Chair — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- center of pulmonary vascular disease, Fuwai hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No